CLINICAL TRIAL: NCT05601167
Title: Open Multicentre Study for Assessment of the Safety and Efficacy Against COVID-19 of the Drug JTBC00201 (PROMOMED RUS LLC, Russia) in the Adult Population
Brief Title: Open Multicentre Study of the Safety and Efficacy Against COVID-19 of Nirmatrelvir/Ritonavir in the Adult Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Promomed, LLC (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NR-012022
Record Dates: First submitted 2022-10-31; First posted 2022-11-01 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: Nirmatrelvir/ritonavir; Skayvira; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JTBC00201 (nirmatrelvir/ritonavir, Skayvira) (Experimental): Group 1 (n=132) received the study drug nirmatrelvir/ritonavir, tablets 300/100 mg, 2 times a day with 12 ±2 hours interval for 5 days in the setting of pathogenetic and symptomatic therapy provided by Interim Guidelines for the prevention, diagnosis and treatment of COVID-19 validated of the time of the study
  Interventions: Drug: nirmatrelvir/ritonavir
- Standard of care (Active Comparator): Group 2 (n=132) patients receive standard therapy prescribed in accordance with the recommended treatment regimens included in the Interim Guidelines for the prevention, diagnosis and treatment of COVID-19 validated of the time of the study
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: nirmatrelvir/ritonavir — Tablets 300/100mg, 2 times a day with 12 ±2 hours interval for 5 days
  Other Names: JTBC00201
  Arms: JTBC00201 (nirmatrelvir/ritonavir, Skayvira)
Drug: Standard of care — The administration of 'Standard of care' drugs was done according to the regimen recommended in the 'COVID-19 TreatmentGuidelines' validated at the time of the study
  Arms: Standard of care

SUMMARY:
This is open-labe randomized multicenter comparative Phase III study conducted in 11 medical facilities. The objective of the study is to evaluate efficacy and safety of the drug JTBC00201, tablets in the setting of pathogenetic and symptomatic therapy as compared to standard therapy in outpatients with COVID-19.

DETAILED DESCRIPTION:
Upon signing the informed consent form and screening, 264 eligible outpatients with mild or moderate COVID-19 were randomized at a 1:1 ratio to receive either nirmatrelvir/ritonavir tablets, 300/100 mg, 2 times a day with 12 ±2 hours interval for 5 days, or SOC

ELIGIBILITY:
Inclusion Criteria:

* Availability of PIS Informed Consent Form signed and dated by a patient.
* Male and female subjects aged 18 to 80 inclusive as of the time of signing the PIS Informed Consent Form.
* Confirmed COVID-19 at screening stage: positive for SARS-CoV-2 RNA laboratory test with nucleic acid amplification techniques (NAAT) or SARS-CoV-2 antigen with immunochromatographic assay.
* SARS-CoV-2 test results obtained up to 5 days prior to randomization may be taken into account upon availability of supporting documentation.
* Mild or moderate SARS-CoV-2 induced infection.
* At least one of the following COVID-19 symptoms as of the time of screening and randomization: nasal congestion or rhinitis; sore throat; dyspnoea or respiratory distress on exertion; cough; tiredness; pain in muscles or throughout the body; headache; chills; fever (body temperature > 38 ⁰С); nausea; vomiting; diarrhoea; anosmia; ageusia.
* Disease onset (first symptom) within not more than 5 days prior to randomization
* The patient agrees and is able to take oral drug products.
* Patient's consent to use reliable contraception methods during the entire study and for 3 weeks after the end of the study. Reliable contraception methods are: sexual abstinence, the use of a condom combined with a spermicidal agent.
* Female subjects incapable of bearing children (history: hysterectomy, tubal ligation, infertility, menopause for more than 2 years), as well as male subjects with infertility or a history of vasectomy may participate in the study.

Exclusion Criteria:

* Hypersensitivity to the study drug components.
* Lactase deficiency, lactose intolerance, glucose-galactose malabsorption.
* Use of direct-acting antiviral drugs within 10 days prior to screening.
* The use of drugs at the time of screening whose clearance is highly dependent on the CYP3A isoenzyme, or which are strong inducers of CYP3A (for more information, see the section "Unauthorized pharmaceuticals").
* Necessity to use unauthorized pharmaceuticals.
* The need for oxygen therapy at the time of screening.
* Hospitalization required at time of screening, or hospitalization expected to be required for COVID-19 within 48 hours of randomization, excluding hospitalization to the observation facility for social reasons (e. g., living in a hostel, cohabiting with people, including those with risk factors for aggravated COVID-19, who, after contact with the patient, have a negative result for the SARS-CoV-2 RNA/antigen, etc.).
* Severe and extremely severe disease signs as of the time of screening.
* Vaccination within less than 4 weeks prior to screening.
* Possible or confirmed moderate COVID-19 within 6 months prior to screening.
* Possible or confirmed history of severe or very severe COVID-19.
* Patients with moderate to severe renal insufficiency (estimated glomerular filtration rate (GFR) < 60 ml/min/1.73 m2 per CKD-EPI formula) or receiving renal replacement therapy at the time of screening.
* Severe liver failure (class C per Child-Pugh) at the time of screening or elevated ALT and/or AST levels of ≥ 2.5 UNL and/or elevated total bilirubin levels of ≥ 2 UNL (≥ 3 UNL with Gilbert's syndrome) in past medical history (within 6 months prior to screening).
* Positive test result for HIV, syphilis, hepatitis B and/or C at the time of screening.
* Alcohol, pharmacological and/or drug dependence (history and/or at the time of screening).
* Schizophrenia, schizoaffective disorder, bipolar disorder, or other psychiatric disorder (history or suspected) at the time of screening.
* Any history data that may complicate, in the opinion of the investigator, interpretation of the study results or create additional risk for the patient due to his/her participation in the study.
* Unwillingness or inability of a patient to comply with the Protocol procedures (in the opinion of the investigator).
* Pregnant or lactating women, or women planning a pregnancy.
* Participation in another clinical study within 3 months prior to enrolment in the present study.
* Other conditions that prevent the patient from inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of patients with COVID-19 severity increase as compared from baseline to Visit 4 | From baseline to Visit 4 (days 14-15)
  Patient severity score at screening and during treatment was determined as per сurrent clinical Guidelines

SECONDARY OUTCOMES:
Clinical status changes according to the WHO Ordinal Scale ranges from 0 (uninfected) to 8 (dead) | From baseline to Visit 2 (days 6-7), 3 (days 11-12), 4 (days 14-15), 5 (days 21±1), 6 (study completion, day 28±1)
  The score as per the categorical ordinal clinical improvement WHO scale
Clinical status deterioration incidence according to the WHO Ordinal Scale ranges from 0 (uninfected) to 8 (dead) by ≥ 1 category | From baseline to Visit 2 (days 6-7), 3 (days 11-12), 4 (days 14-15)
  The proportion of patients with clinical status deterioration as per the categorical ordinal clinical improvement on the WHO scale of ≥1 category
Achievement of clinical status 0 according to the WHO Ordinal Scale ranges from 0 (uninfected) to 8 (dead) | From baseline to Visit 2 (days 6-7), 3 (days 11-12), 4 (days 14-15)
  The proportion of patients with category 0 as per the categorical ordinal clinical improvement on the WHO scale
Prevalence of patients with negative SARS-CoV-2 RNA test | From baseline to Visit 2 (days 6-7), 3 (days 11-12), 4 (days 14-15)
  The proportion of patients with negative SARS-CoV-2 RNA test
Symptoms intensity score as per COVID-19 Related Symptom Scale | From baseline to Visit 2 (days 6-7), 3 (days 11-12), 4 (days 14-15), 5 (days 21±1), 6 (study completion, day 28±1)
  The proportion of patients with Symptoms intensity score as per COVID-19 Major Symptom Rating Scale. Ranges for each symptom: 0 points (no symptoms) - 3 points (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy Pushkar, Academician, Principal Investigator — Moscow State Clinical Hospital №50
Locations (11):
- Russia (11):
  - Regional Budgetary Healthcare Institution "Ivanovo Clinical Hospital", Ivanovo
  - Kirov State Medical University of Ministry of Health of the Russian Federation, Kirov
  - State Budgetary Healthcare Institution City Clinical Hospital named after S. I. Spasokukotskiy of Moscow Healthcare Department, Moscow
  - Regional Clinic Hospital of Ryazan, Ryazan
  - Ryazan State Medical University named after academician I.P. Pavlov of Ministry of Health of the Russian Federation, Ryazan
  - Avrora MedFort, LLC, Saint Petersburg
  - OrCli Hospital, LLC, Saint Petersburg
  - Ogarev Mordova State University of Ministry of Health of the Russian Federation, Saransk
  - Regional State Budgetary Healthcare Institution "Clinical Hospital No. 1", Smolensk
  - Smolensk State Medical University of Ministry of Health of the Russian Federation, Smolensk
  - State Budgetary Healthcare Institution of the Yaroslavl Oblast "Clinical Hospital No.3", Yaroslavl

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] L.A. Balykova, N.M. Selezneva, E.I. Gorshenina, O.I. Shepeleva, N.V. Kirichenko, E.N. Simakina, K.B. Kolontarev, D.Yu. Pushkar, D.N. Zemskov, K.Ya. Zaslavskaya, S.M. Noskov, A.V. Taganov, P.A. Bely. modern directed antiviral COVID-19 therapy: results of multicenter clinical effectiveness and safety study of fixed nirmatrelvir+ritonavir combination. Pharmacy & Pharmacology. 2022;10(4):. DOI: 10.19163/2307-9266- 2022-10-4-
- See also: Cyberleninka is an open access scientific electronic library — https://cyberleninka.ru/article/n/sovremennaya-napravlennaya-protivovirusnaya-terapiya-covid-19-rezultaty-mnogotsentrovogo-klinicheskogo-issledovaniya-effektivnosti